CLINICAL TRIAL: NCT01107665
Title: A Phase II, Single-Arm Study of Pazopanib and Paclitaxel as First-Line Treatment for Subjects With Unresectable Stage III and Stage IV Melanoma
Brief Title: Pazopanib and Paclitaxel as First-Line Treatment for Subjects With Unresectable Stage III and Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, John P. Fruehauf, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 09-53; 2010-7443 (Other: University of California, Irvine); PZP113567 (Other: GlaxoSmithKline); NCI-2010-00748 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Stage III Melanoma; Stage IV Melanoma; Unresectable Melanoma
Keywords: pazopanib; paclitaxel; melanoma
MeSH Terms: conditions — Melanoma | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib and Paclitaxel (Experimental): Treatment on study will be administered in 4-week cycles. Paclitaxel will be administered intravenously at a starting dose of 80mg/m2 weekly for 3 weeks followed by a 1-week rest. Pazopanib will be administered orally, in a continuous regimen, with a starting dose of 800mg daily.
  Interventions: Drug: Pazopanib and Paclitaxel

INTERVENTIONS:
Drug: Pazopanib and Paclitaxel — Paclitaxel will be administered intravenously at a starting dose of 80mg/m2 weekly for 3 weeks followed by a 1-week rest. Pazopanib will be administered orally, in a continuous regimen, with a starting dose of 800mg daily.
  Other Names: Pazopanib monohydrochloride salt and Taxol

SUMMARY:
This is a Phase II single-arm, open-label, clinical trial evaluating the efficacy and safety of pazopanib in combination with paclitaxel as first line therapy for subjects with unresectable Stage III and Stage IV melanoma. Previous cytokine therapy is permitted. Subjects must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST). Subjects who are not candidates for curative intent treatments are eligible for this study.

DETAILED DESCRIPTION:
Treatment on study will be administered in 4-week cycles. Paclitaxel will be administered intravenously at a starting dose of 80mg/m2 weekly for 3 weeks followed by a 1-week rest. Pazopanib will be administered orally, in a continuous regimen, with a starting dose of 800mg daily.

Approximately 60 eligible subjects will be enrolled over a 24 month period. 21 subjects will be entered into the first stage of a 2-stage Simon Minimax design. If there are 3 or more responses, 39 additional subjects will be enrolled in Stage 2. The minimum number of responses required to move to the second stage, > 3, were noted after the first 9 patients on treatment, and the study then proceeded towards the goal of accruing 60 total patients. Subjects are permitted to receive supportive care throughout the study including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrheal agents, analgesics, erythropoietin, filgrastim (Neupogen), or bisphosphonates, when appropriate. Subjects should continue treatment on study until objective disease progression is documented according to RECIST or withdrawal from the study for other reasons. Subjects discontinuing treatment with paclitaxel prior to disease progression should continue treatment with pazopanib. Subjects discontinuing both agents prior to progressive disease (PD) will be followed for tumor assessment until PD, or until the initiation of a subsequent anti-cancer therapy in the absence of documented PD, or until death, whichever occurs first. Subjects may continue treatment beyond the time of RECIST-defined progression at the discretion of the investigator if the subject is perceived to be experiencing clinical benefit. Overall survival will be assessed for 2 years from first study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol. Note: It is not necessary that informed consent be obtained within the protocol-specified screening window.
2. Histologically confirmed cutaneous melanoma with 1) unresectable Stage III disease, or 2) Stage IV disease by American Joint Committee on Cancer (AJCC) criteria.
3. Must have measurable disease [i.e. with at least one measurable lesion, per RECIST]. A measurable lesion is defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥20mm using conventional techniques or ≥10mm with spiral CT scan.

   Note: Subjects should be excluded if all baseline measurable lesions are within previously irradiated areas. Subjects participating in the exploratory analysis shall not have the biopsied lesion(s) as the only sites of measurable disease.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Age 18 years old or older
6. A female is eligible to enter and participate in this study if she is of:

   Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
   * A hysterectomy
   * A bilateral oophorectomy (ovariectomy)
   * A bilateral tubal ligation
   * Is post-menopausal

   Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 milliinternational unit (mIU)/mL and an estradiol value <40pg/mL (<140 pmol/L).

   Subjects must discontinue HRT prior to study enrollment due to the potential for inhibition of Cytochrome P450 (CYP) enzymes that metabolize estrogens and progestins. For most forms of HRT, at least 2-4 weeks must elapse between the cessation of HRT and determination of menopausal status; length of this interval depends on the type and dosage of HRT. If a female subject is determined not to be post-menopausal, they must use adequate contraception, as defined immediately below.

   Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
   * An intrauterine device with a documented failure rate of less than 1% per year.
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
   * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

   Note: Oral contraceptives are not reliable due to potential drug drug interactions.

   Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

   A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.
7. Adequate organ system functions as defined below:

   System:Laboratory Values

   Hematologic
   * Absolute neutrophil count (ANC) >= .5 X 10^9/L
   * Hemoglobin >= 9 g/dL
   * International normalized ratio (INR) <= 1.2 X upper limit of normal (ULN)
   * Partial thromboplastin time (PTT) <= 1.2 X ULN

   Hepatic
   * Total bilirubin <= 1.5 X ULN
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <=2.5 x ULN

   Renal
   * Calculated creatinine clearance >= 30 mL/min Note: Subjects may not have had a transfusion within 7 days of screening assessment.
   * Platelets >= 100 X 10^9/L
   * Urine Protein to Creatinine Ratio (UPC) < 1 Note: If UPC is more than 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1g to be eligible.
8. Corrected serum calcium concentration within normal range per local clinical laboratory standard.
9. Left ventricular ejection fraction (LVEF) more or equal lower limit of normal (LLN) as assessed by echocardiography or multigated acquisition (MUGA) scan.

Exclusion Criteria:

* Subjects meeting any of the following criteria must not be enrolled in the study:

  1. Prior treatment with cytotoxic anti-cancer therapy. (Previous cytokine or investigational immunotherapy are permitted, but must be completed 28 days prior to first dose of study medication).
  2. Prior use of other investigational or licensed tyrosine kinase inhibitors (TKIs), or agents which target vascular endothelial growth factor (VEGF) or VEGF receptors (ie. bevacizumab, VEGF-Trap).
  3. Known history of dose-limiting hypersensitivity reactions to paclitaxel/Cremophor EL.
  4. Pregnant or lactating female. Female subjects who are lactating are eligible if they discontinue nursing prior to the first dose of study drug and refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
  5. Melanoma of ocular origin.
  6. History of another malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
  7. Life expectancy less than 3 months.
  8. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis except for subjects who have previously-treated CNS metastases (surgery with or without radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria:

     1. Are asymptomatic
     2. Have had no evidence of active CNS metastases for more or equal 6 months prior to enrollment
     3. Have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC)
  9. Clinically significant gastrointestinal abnormalities including, but not limited to:

     1. Malabsorption syndrome
     2. Major resection of the stomach or small bowel that could affect the absorption of study drug
     3. Active peptic ulcer disease
     4. Inflammatory bowel disease
     5. Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
     6. History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
  10. Presence of uncontrolled infection.
  11. Prolongation of corrected QT interval (QTc) >480 milliseconds (ms).
  12. History of any one or more of the following cardiovascular conditions within the past 6 months:

      1. Cardiac angioplasty or stenting
      2. Myocardial infarction
      3. Unstable angina
      4. Symptomatic peripheral vascular disease
      5. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
  13. History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
  14. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥150 millimeters of mercury (mmHg)or diastolic blood pressure (DBP) of ≥ 90 mmHg].

      Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP/DBP values from each blood pressure assessment must be less or equal 150 systolic and 90 diastolic mmHg in order for a subject to be eligible for the study.
  15. Prior major surgery or trauma within 14 days of the first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
  16. Evidence of active bleeding or bleeding diathesis
  17. Hemoptysis within 6 weeks of first dose of study drug.
  18. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.
  19. Use of any prohibited medications within 14 days of the first dose of study medication.
  20. Radiation therapy within 28 days of the first dose of study drug.
  21. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity.
  22. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fruehauf, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- [Result] Fruehauf JP, El-Masry M, Osann K, Parmakhtiar B, Yamamoto M, Jakowatz JG. Phase II study of pazopanib in combination with paclitaxel in patients with metastatic melanoma. Cancer Chemother Pharmacol. 2018 Aug;82(2):353-360. doi: 10.1007/s00280-018-3624-6. Epub 2018 Jun 25. PMID 29943192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazopanib and Paclitaxel
Started | 60
Completed (Subjects who completed protocol-defined follow-up period.) | 11
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival at 6 Months
Description: This is defined as the percentage of subjects who are free of RECIST-defined objective disease progression at 6 months after study treatment start. Subjects in the Intent-to-Treat (ITT) population who discontinue the study prior to 6 months will be included in the denominator when calculating the percentage. Progression is defined using the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 68

2. Secondary Outcome: Percentage of Participants Alive at 1 Year
Description: This is defined as the percentage of subjects who are alive at 1 year after enrollment. For subjects who do not die, time to death will be censored at the time of last contact.
Time Frame: At 1 year after enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 48

3. Secondary Outcome: Percentage of Participants Alive at 2 Years
Description: This is defined as the percentage of subjects who are alive at 2 years after enrollment. For subjects who do not die, time to death will be censored at the time of last contact.
Time Frame: At 2 years after enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 27

4. Secondary Outcome: Objective Response Rate (ORR)
Description: This is defined as the percentage of subjects achieving either a complete or partial tumor response per RECIST criteria. The response rate will be calculated from the review of best response which records confirmed cases of PR and CR only. Confirmation will occur at least 4 weeks after the initial response. Stable disease (SD) will also be defined by 8 weeks or greater and will be summarized by less than 6 months vs. equal or greater than 6 months. Subjects in the ITT population with unknown or missing response will be treated as non-responders, i.e. they will be included in the denominator when calculating the percentage. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of the longest diameter of target lesions; Overall Reponse (ORR) = CR + PR.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 36

5. Secondary Outcome: Clinical Benefit Response (CBR)
Description: This is defined as the percentage of subjects achieving either a complete (CR), partial tumor (PR) or stable disease (SD) response per RECIST criteria. Confirmation will occur at least 4 weeks after the initial response for partial and complete responders. Stable disease will also be defined by 8 weeks or greater.
  Subjects in the ITT population with unknown or missing response will be treated as non-responders, i.e. they will be included in the denominator when calculating the percentage. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD or the persistence of one ore more non-target lesions; Clinical Benefit Rate = (SD+PR+CR).
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 91

6. Secondary Outcome: Duration of Response (DR)
Description: Duration of response analyses will be restricted to the subgroup of the population who experience a response during the study. Duration of response will be defined as the time from first documented evidence of response (CR/PR) until the first documented sign of disease progression or death, if sooner. For subjects who do not progress or die, duration of response will be censored on the date of last assessment.
  Duration of response will be summarized using the Kaplan-Meier method.
Time Frame: Time from first documented evidence of response (CR/PR) until the first documented sign of disease progression or death, assessed up to 2 years
Population: Duration of response analyses will be restricted to the subgroup of the population who experience a response during the study. Duration of response will be defined as the time from first documented evidence of response (CR/PR) until the first documented sign of disease progression or death, if sooner.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 20
days | 351.7 (284.9)

7. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Safety Parameters
Description: AEs and toxicities will be graded according to the National Cancer Institute-common toxicity criteria (NCI-CTC), Version 3.0. Summaries of the number of toxicity grades for both laboratory and non-laboratory data will be presented. If the AE is listed in the NCI-CTC, the maximum grade will be summarized. Otherwise, the maximum intensity will be summarized. AEs will be coded using the standard dictionary (MedDRA), and grouped by system organ class. They will be summarized by frequency and proportion of total subjects, by system organ class and preferred term. Separate summaries will be given for all AEs, for drug-related AEs, for SAEs, and for AEs leading to withdrawal from the study treatment. The incidence of deaths will also be reported.
  Please refer to the Adverse Event table for specifics.
Time Frame: From baseline until date of first documented progression, until initiation of a subsequent anti-cancer therapy, until death, whichever came first, assessed until death, the patient withdraws consent, or the study ends, up to 2 years
Population: Please refer to the Adverse Event tables for specifics.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 60
Participants | 60

8. Other Pre Specified Outcome: Concentrations of Plasma Proteins (Serum VEGF, Soluble VEGF Receptor 2, Serum Hypoxia-inducible Factor (HIF) and Serum TSP1) That May be Associated to Angiogenesis and Tumor Proliferation
Description: Categorical statistical analysis will be performed to determine the relationship between PD and pharmacokinetic (PK) markers and outcomes. Univariate summary statistics will be calculated, such as the sample median, standard deviation, minimum, and maximum observations. The dichotomized variables were tabulated as high and low levels or positive and negative expression. Changes over time in continuously distributed biomarker levels will be investigated with the sign's test because of the heavy degree of skewness observed in some of the marginal distributions. There are no results for this exploratory endpoint due to cuts in funding.
Time Frame: Day 1
Population: Exploratory endpoints were not analyzed due to depletion of funds.
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Tissue Levels of Angiogenic Markers Including Protein (p)53, HIF, Cluster of Differentiation (CD)31, Neuronal Nitric Oxide Synthase (nNOS), TSP1, and VEGF
Description: Categorical statistical analysis will be performed to determine the relationship between PD and PK markers and outcomes. Univariate summary statistics will be calculated, such as the sample median, standard deviation, minimum, and maximum observations. The dichotomized variables were tabulated as high and low levels or positive and negative expression. Changes over time in continuously distributed biomarker levels will be investigated with the sign's test because of the heavy degree of skewness observed in some of the marginal distributions. There are no results for this exploratory endpoint due to cuts in funding.
Time Frame: Day 1
Population: Exploratory endpoints were not analyzed due to depletion of funds.
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: In Vitro Response of Tumor Cells Grown in Culture With Vascular Endothelial Cells to Pazopanib, Paclitaxel, Topotecan and Resveratrol
Description: In vitro response of tumor cells grown in culture with vascular endothelial cells to pazopanib, paclitaxel, topotecan and resveratrol. There are no results for this exploratory endpoint due to cuts in funding.
Time Frame: Day 1
Population: Exploratory endpoints were not analyzed due to depletion of funds.
Arm/Group | Pazopanib and Paclitaxel
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: (BRAF) Mutation Status vs Survival
Description: Comparison of OS between BRAF mutant subset and BRAF WT/unknown group.
Time Frame: Up to 36 months
Population: Stage III/IV melanoma
Measure: Median (95% Confidence Interval); unit: months
Groups:
- BRAF Mutant Subset: Subset of subjects who are BRAF mutant positive
- BRAF WT/Unknown Group: Subset of subjects who are BRAF WT or unknown status.
Arm/Group | BRAF Mutant Subset | BRAF WT/Unknown Group
Number analyzed (Participants) | 14 | 46
months | 18 [12.6 to 22.6] | 11.3 [8 to 13.5]
Statistical Analysis 1: Comparison: BRAF Mutant Subset vs BRAF WT/Unknown Group; Test type: Other; p = 0.49, Log Rank; Log Rank HR = 0.784, 95% CI 2-sided [.41 to 1.54]

ADVERSE EVENTS:
Time Frame: Adverse events were collected and recorded from receipt of first receipt of first of study drug until 28 days have elapsed following cessation of study drug, regardless of initiation of a new cancer therapy or transfer to hospice.
Description: AEs were collected systematically through regular investigator assessments and laboratory testing.
  SAEs were either grade 3 or 4 according to the NCI Common Terminology Criteria for Adverse Events, version 3.0.
Arm/Group | Pazopanib and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 10/60
Other Adverse Events (participants affected / at risk) | 44/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib and Paclitaxel (N=60)
Fatigue (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 3
Hypertension (Cardiac disorders) | 1
Transaminitis (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 9
Nausea (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib and Paclitaxel (N=60)
Fatigue (General disorders) | 44
Diarrhea (Gastrointestinal disorders) | 37
Hypertension (Cardiac disorders) | 35
Nausea (General disorders) | 29
Transaminitis (Blood and lymphatic system disorders) | 21
Anemia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 18

LIMITATIONS AND CAVEATS:
Analysis on one secondary outcome and other exploratory outcomes were not performed due to depleted funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT01107665/Prot_SAP_000.pdf